CLINICAL TRIAL: NCT07335562
Title: A Phase 3, Randomized, Open-label, Multicenter Study to Compare the Efficacy and Safety of BMS-986353, CD19-targeted NEX-T CAR T Cells, Versus Standard of Care in Participants With Active Systemic Sclerosis (Breakfree-SSc)
Brief Title: A Study to Compare the Efficacy and Safety of BMS-986353 (Zolacaptagene- Autoleucel / Zola-cel), CD19-CAR T Cells, Versus Standard of Care in Participants With Active Systemic Sclerosis
Acronym: Breakfree-SSc
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Juno Therapeutics, Inc., a Bristol-Myers Squibb Company (Industry)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA061-1005; 2025-524337-11 (Other: EU CT Number); U1111-1330-3381 (Other: UTN)
Record Dates: First submitted 2026-01-09; First posted 2026-01-13 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Systemic | interventions — fludarabine; Cyclophosphamide; tocilizumab; Rituximab; nintedanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: BMS-986353 (Experimental)
  Interventions: Drug: BMS-986353; Drug: Fludarabine; Drug: Cyclophosphamide
- Arm B: Standard of Care (Experimental)
  Interventions: Drug: Tocilizumab; Drug: Rituximab; Drug: Nintedanib

INTERVENTIONS:
Drug: BMS-986353 — Specified dose on specified days
  Other Names: CC-97540
  Arms: Arm A: BMS-986353
Drug: Fludarabine — Specified dose on specified days
  Arms: Arm A: BMS-986353
Drug: Cyclophosphamide — Specified dose on specified days
  Arms: Arm A: BMS-986353
Drug: Tocilizumab — Specified dose on specified days
  Arms: Arm B: Standard of Care
Drug: Rituximab — Specified dose on specified days
  Arms: Arm B: Standard of Care
Drug: Nintedanib — Specified dose on specified days
  Arms: Arm B: Standard of Care

SUMMARY:
The purpose of this study is to compare the efficacy and safety of BMS-986353 versus standard of care in participants with active Systemic Sclerosis

ELIGIBILITY:
Inclusion Criteria

- Participants must fulfill the 2013 American College of Rheumatology (ACR) / European League Against Rheumatism (EULAR) classification criteria for Systemic Sclerosis (SSc), and additionally have the following:.

i) Positive Antinuclear Antibodies (ANA) with nucleolar pattern and/or anti-Topoisomerase I (anti-Scl-70) antibodies.

ii) Confirmation of Interstitial Lung Disease (ILD) on centrally read High-Resolution Computed Tomography (HRCT) with ≥ 10% total lung involvement, with at least one of the following attributed to active SSc:.

A. Arthritis.

B. Myositis.

C. Carditis.

D. Progressive skin disease.

E. Elevated inflammatory markers.

- Participants must have a non-response or intolerance despite ≥ 6 months of treatment with at least one immunomodulatory drug. Non-response is defined as a patient, who in the opinion of the investigator, is not adequately controlled/treated and requires treatment escalation.

Exclusion Criteria

* Participants must not have a requirement for supplemental oxygen therapy and/or Diffusing Capacity of the Lungs for Carbon Monoxide (DLCO) ≤ 40% (Hemoglobin (Hgb) corrected) at screening.
* Participants must not have moderate to severe Pulmonary Arterial Hypertension (PAH) requiring PAH-specific combination treatment
* Participants must not have pulmonary comorbidity including chronic obstructive pulmonary disease or asthma requiring daily oral corticosteroids, cigarette smoking (including e-cigarettes) within 3 months before screening or unwilling to avoid smoking throughout the study, and/or clinically significant abnormalities on HRCT not attributable to SSc assessed by the central reader at screening.
* Participants must not have gastrointestinal (GI) dysmotility requiring Total Parenteral Nutrition (TPN).
* Participants must not have current gangrene of a digit
* Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2026-04-30 (Estimated); Primary Completion 2028-11-14 (Estimated); Study Completion 2030-11-11 (Estimated)

PRIMARY OUTCOMES:
The absolute change from baseline in Forced Vital Capacity (FVC) in mL | At 12 months

SECONDARY OUTCOMES:
The absolute change from baseline in Modified Rodnan Skin Score (mRSS) | At month 12
The absolute change from baseline in Quantitative Interstitial Lung Disease-Whole Lung (QILD-WL) score | Up to month 36
Time to progression, defined as the time from randomization to progressive disease | Approximately 54 months
The change from baseline in Patient-Reported Outcomes Measurement Information System (PROMIS)-Fatigue | Up to month 36
The change from baseline in Scleroderma Clinical Index (ScleroID) | Up to month 36
The change from baseline in Scleroderma Health Assessment Questionnaire - Disability Index (SHAQ-DI) | Up to month 36
The change from baseline in PROMIS-29 | Up to month 36
The change from baseline in St. George's Respiratory Questionnaire (SGRQ) | Up to month 36
The change from baseline in EuroQol 5 Dimensions 5 Level (EQ-5D-5L) visual analog scale | Up to month 36
The change from baseline in EQ-5D-5L Utility Index | Up to month 36
The absolute change from baseline in FVC in mL | Up to month 36
The absolute change from baseline in FVC in mL/year | Up to month 36
The absolute change from baseline in Percent Predicted Forced Vital Capacity (ppFVC) | Up to month 36
The relative change from baseline in ppFVC | Up to month 36
The absolute change from baseline in diffusing capacity of the lung for carbon monoxide (DLCO) | Up to month 36

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (51):
- United States (14):
  - Local Institution - 0035, Scottsdale, Arizona
  - Local Institution - 0092, Aurora, Colorado
  - Local Institution - 0001, Denver, Colorado
  - Local Institution - 0069, Miami, Florida
  - Local Institution - 0014, Atlanta, Georgia
  - Local Institution - 0139, Chicago, Illinois
  - Local Institution - 0084, Worcester, Massachusetts
  - Local Institution - 0034, Ann Arbor, Michigan
  - Local Institution - 0037, Rochester, Minnesota
  - Local Institution - 0082, Summit, New Jersey
  - Local Institution - 0122, Cleveland, Ohio
  - Local Institution - 0002, Charleston, South Carolina
  - Local Institution - 0074, Dallas, Texas
  - Local Institution - 0008, Seattle, Washington
- Belgium (3):
  - Local Institution - 0003, Antwerp, Flanders
  - Local Institution - 0057, Leuven, Vlaams-Brabant
  - Local Institution - 0080, Liège
- Canada (2):
  - Local Institution - 0104, Halifax, Nova Scotia
  - Local Institution - 0088, Sherbrooke, Quebec
- France (5):
  - Local Institution - 0031, Strasbourg, Alsace
  - Local Institution - 0061, Toulouse, Haute-Garonne
  - Local Institution - 0049, Bordeaux
  - Local Institution - 0012, Bron
  - Local Institution - 0052, Paris
- Germany (7):
  - Local Institution - 0046, Berlin
  - Local Institution - 0016, Cologne
  - Local Institution - 0028, Erlangen
  - Local Institution - 0042, Leipzig
  - Local Institution - 0032, München
  - Local Institution - 0033, Tübingen
  - Local Institution - 0038, Würzburg
- Italy (4):
  - Local Institution - 0103, Rome, Lazio
  - Local Institution - 0004, Milan, Milano
  - Local Institution - 0108, Pisa, Tuscany
  - Local Institution - 0106, Milan
- Japan (6):
  - Local Institution - 0026, Sapporo, Hokkaido
  - Local Institution - 0132, Yokohama, Kanagawa
  - Local Institution - 0137, Suita, Osaka
  - Local Institution - 0117, Bunkyo-ku, Tokyo
  - Local Institution - 0123, Fukuoka
  - Local Institution - 0118, Okayama
- Spain (4):
  - Local Institution - 0129, A Coruña, A Coruña [La Coruña]
  - Local Institution - 0138, Barcelona, Catalunya [Cataluña]
  - Local Institution - 0060, Barcelona
  - Local Institution - 0009, Málaga
- Switzerland (3):
  - Local Institution - 0047, Basel
  - Local Institution - 0068, Bern
  - Local Institution - 0078, Zurich
- United Kingdom (3):
  - Local Institution - 0063, Leeds, West Yorkshire
  - Local Institution - 0091, Sheffield, Yorkshire and the Humber
  - Local Institution - 0059, London

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT07335562.html